CLINICAL TRIAL: NCT03803124
Title: Effect of Tolvaptan on Renal Plasma Flow (RPF) and Glomerular Filtration Rate (GFR) in ADPKD
Acronym: POLY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FHM-1-2015
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: CYSTS, KIDNEYS
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Cysts | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan (Active Comparator): Drug: Tolvaptan
  1 tablet before renography
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Placebo
  1 tablet before renography
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — 1 tablet before renography
  Arms: Tolvaptan
Drug: Placebo — 1 tablet before renography
  Arms: Placebo

SUMMARY:
Polycystic kidney disease (ADPKD) is a common genetic disorder, characterized by the formation of cysts in the kidneys, causing gradual renal function-loss. Previous studies have shown that, reduced glomerular filtration rate (GFR) and renal plasma flow (RPF) play a role in the progression of renal disease in ADPKD. Tolvaptan is a vasopressin 2 antagonist, which seems to reduce the growth of total kidney volume (TKV) and the decline in e-GFR in ADPKD. The mechanism is not fully understood and could, at least partly, be caused by stimulation of the renal blood flow. The purpose of this trial is to investigate if tolvaptan´s improve renal blood flow and glomerular filtration in ADPKD, in a randomized, cross-over, double-blind, placebo-controlled study.

DETAILED DESCRIPTION:
The aim is to measure the acute effects of tolvaptan on:

1. Renal hemodynamics (RPF, GFR, filtration fraction ((FF)) and renovascular resistance ((RVR))
2. Blood pressure (central blood pressure ((cBP)) and brachial blood pressure bBP)
3. Several vasoactive hormones (plasma renin ((PRC)), plasma angiotensin II ((p-Ang-II)), plasma aldosterone ((p-Aldo)), plasma vasopressin ((p-AVP))

in patients with ADPKD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis with ADPKD
* Informed consent
* Contraception for fertile women

Exclusion Criteria:

* Renal transplantation
* Operation in the kidney
* Diabetes mellitus
* Neoplastic conditions
* Pregnancy, nursing
* Unwillingness to participate
* eGFR > 30
* Intolerance towards tolvaptan
* Alcohol or medical abuse,
* BP >>170/110 blood pressure despite regulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Renal plasma flow (RPF) | Two hours after trial medicine intake
  Estimated by posterior Technetium-99m diethylenetriamine penta-acetic acid (99-mTc-DTPA) renography 2 hours after trial medicine intake. (unit of measurement= ml/min)

SECONDARY OUTCOMES:
Central and brachial blood pressures (BP) | Measured every 15 minutes during the examination day
  Measured using Mobil-O-Graph® PWA (unit of measurement= mmHg)
Glomerular filtration rate (GFR) | Two hours after trial medicine intake
  Estimated by posterior Technetium-99m diethylenetriamine penta-acetic acid (99-mTc-DTPA) renography 2 hours after trial medicine intake. (unit of measurement= ml/min)
Filtration fraction (FF) | Two hours after trial medicine intake
  Estimated by posterior Technetium-99m diethylenetriamine penta-acetic acid (99-mTc-DTPA) renography 2 hours after trial medicine intake. (unit of measurement= %)
Plasma concentration of vasopressin (p-AVP) | Measured before and 3 hours after trial medicine intake
  Blood samples (unit of measurement= pg/ml)
Plasma concentration of aldosterone (p-Aldo) | Measured before and 3 hours after trial medicine intake
  Blood samples (unit of measurement= pmol/ml)
Plasma concentration of angiotensin II (p-AngII) | Measured before and 3 hours after trial medicine intake
  Blood samples (unit of measurement= pg/ml)
Plasma concentration of renin (PRC) | Measured before and 3 hours after trial medicine intake
  Blood samples (unit of measurement= pg/ml)
Urine excretion of aquaporin 2 (u-AQP2) | Measured before and 3 hours after trial medicine intake
  Urine sample (unit of measurement= ng/ml)
Urine output (OU) | Measured before and 3 hours after trial medicine intake
  Urine sample (unit of measurement= ml/min)
Urine osmolality (U-osm) | measured before and 3 hours after trial medicine intake
  Urine sample (unit of measurement= mosmol/kg)
Fractional excretion of sodium (FENa) | Measured before and 3 hours after trial medicine intake
  Blood and urine sample (unit of measurement= %)
Albumin excretion rate | Measured before and 3 hours after trial medicine intake
  Blood and urine sample (unit of measurement= mg/min)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Mose, MD, Ph D, Principal Investigator — Departments of medical research and medicine
Locations (1):
- Departments of medical research and medicine, Holstebro, Denmark